CLINICAL TRIAL: NCT05448196
Title: Assessing the Impact of a Financial Navigation Program for Patients With Multiple Myeloma: a Randomized Controlled Trial
Brief Title: Assessing the Impact of a Financial Navigation Program for Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 39421; 850241 (Other: Penn Medicine)
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Financial Toxicity
MeSH Terms: conditions — Multiple Myeloma; Financial Stress

STUDY DESIGN:
Intervention Model Description: Patients who consent to participation will complete an 11-item screener (the COST22; see "Primary Outcome" and "Screener"). Participants who are not at risk of financial toxicity (COST score ≥26) will be followed longitudinally (i.e., they will be given baseline and 4-month follow up assessments). Patients who score <26 will be identified as being at risk of financial hardship and will be eligible for randomization to a coordinated financial navigation program or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to the intervention arm will be enrolled in a four-month coordinated financial navigation program. This program will take a more proactive, coordinated, and systematic approach and includes concrete action plans, and frequent and standardized follow-ups. All patients randomized to the intervention arm will meet with the nurse navigator (NN) for an intake. The NN will introduce navigation services and navigator's NN role and describe the financial navigation program (e.g., goals and expectations of the financial advocacy and social work programs). Next, the navigator will elicit from the patient their potential and current barriers to completing the diagnostic test or treatment. The navigator will then perform proactive outreach to these resources and coordinate an action plan with the patient.
  Interventions: Other: Coordinated Financial Navigation Program
- Usual Care (No Intervention): Patients are connected to financial advocacy and social work on an ad hoc basis, rather than systematically. We hypothesize that many patients who would qualify and benefit from these services are not using them or are being referred late in their treatment course, which is contributing to their financial hardship and adversely affecting their healthcare.

INTERVENTIONS:
Other: Coordinated Financial Navigation Program — Patients randomized to the intervention arm will be enrolled in a four-month coordinated financial navigation program. This program will take a more proactive, coordinated, and systematic approach and includes concrete action plans, and frequent and standardized follow-ups. All patients randomized to the intervention arm will meet with the nurse navigator (NN) for an intake. The NN will introduce navigation services and navigator's NN role and describe the financial navigation program (e.g., goals and expectations of the financial advocacy and social work programs). Next, the navigator will elicit from the patient their potential and current barriers to completing the diagnostic test or treatment. The navigator will then perform proactive outreach to these resources and coordinate an action plan with the patient.
  Arms: Intervention

SUMMARY:
The study is a randomized controlled trial to develop and evaluate a coordinated financial navigation program at the Abramson Cancer Center (ACC) for patients with multiple myeloma and identify barriers to its broader implementation.

DETAILED DESCRIPTION:
Many financial support services are available to patients at the ACC, but are offered by different umbrella departments and rely on self- or clinician-referrals. Financial Advocacy provides assistance with insurance benefits, copayment assistance and hospital-based financial support. Social work assists with costs not directly related to treatment and also connects patients with community resources. Programs that increase coordination between these departments and proactively screen patients for financial hardship may enhance the reach of available services. However, such programs are resource intensive. As such, obtaining a better understanding of their benefits and any barriers to their expansion is a necessary first step to their broader implementation.

The long-term goal is to implement evidence-based practices that reduce ACC patients' financial burden. The overall objective of this proposal is to develop and evaluate a coordinated financial navigation program at the ACC for patients with multiple myeloma and identify barriers to its broader implementation. The rationale is that understanding the program's effectiveness and any barriers to its scalability will guide the way in which it could be incorporated into existing ACC workflows to maximize benefit for patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients actively receiving systemic therapy at the ACC, defined as receiving any anti-myeloma treatment and at least monthly follow-up at PCAM4 or one of our satellite locations (CCH, Princeton, Lancaster, Cherry Hill, Valley Forge, Radnor)

  * These patients will be approached/recruited in-person on the same date as their return visit (follow-up appointment for established patients)
  * These patients may have already been seen by FA/SW (we will record this information and control for this in the final statistical models)
  * The rationale for using the "follow up at least monthly" criterion is because it will allow our research coordinators to easily and readily review charts of patients scheduled for follow up with myeloma specialists. This strategy will only exclude patients who receive oral maintenance anti-myeloma therapy who follow up less than once monthly (e.g. lenalidomide maintenance only).

    2. New patients expected to start therapy, who are expected to meet criterion #1.
  * These patients will be approached/recruited at their first return visit.
  * If these patients are not expected to return within 2 weeks of the initial visit, a telephone consent will be considered/offered

Exclusion Criteria:

* o Have completed induction treatment and have stopped all systemic treatment in preparation for an autologous stem cell transplant [SCT] (rationale: patients are pre-screened for being able to finance their transplant before proceeding)

  * Are referred only for autologous SCT (they would not qualify by criterion #1, anyway)
  * Actively receive systemic therapy but do not follow up more than once monthly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
COmprehensive Score for Financial Toxicity (COST) | 4 months
  Primary outcome is assessing for change in participants' COmprehensive Score for Financial Toxicity (COST) from the baseline assessment to repeat assessment after 4 months of financial navigation. Scores range from 0-44, with lower scores representing greater financial hardship.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy (FACT-G) | 4 months
  Secondary outcome is assessing for change in participants' Health Related Quality of Life (HRQOL) as measured in part by the Functional Assessment of Cancer Therapy (FACT-G) from the baseline assessment to repeat assessment after 4 months of financial navigation. The FACT-G includes 4 subscales (physical well-being, social/family well-being, emotional well-being, and functional well-being). The score ranges from 0-108 with a higher score indicating better quality of life.
Patient Satisfaction Questionnaire Short-Form [PSQ-18] | 4 months
  Secondary outcome is assessing for change in participants' HRQOL as measured in part by the Patient Satisfaction Questionnaire Short-Form [PSQ-18] from the baseline assessment to repeat assessment after 4 months of financial navigation. The PSQ-18 includes 7 subscales (general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and convenience). The score ranges from 18-90 points with higher scores indicating increased patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Stadtmauer, MD, Principal Investigator — Penn Medicine
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided